CLINICAL TRIAL: NCT00003649
Title: Phase I Pilot Trial of Adenovirus p53 in Bronchioloalveolar Cell Lung Carcinoma (BAC) Administered by Bronchoalveolar Lavage
Brief Title: Gene Therapy in Treating Patients With Non-small Cell Lung Cancer That Cannot Be Surgically Removed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066741; E-6597
Record Dates: First submitted 1999-11-01; First posted 2003-04-30 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — advexin

INTERVENTIONS:
Biological: Ad5CMV-p53 gene

SUMMARY:
RATIONALE: Exposing tumor cells to the p53 gene may improve the body's ability to fight non-small cell lung cancer.

PURPOSE: Phase I trial to study the effectiveness of gene therapy in treating patients who have non-small cell lung cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety of multiple endobronchial treatments with adenovirus p53 bronchoalveolar lavage of a single lobe of the lung in patients with bronchoalveolar cell lung carcinoma.
* Evaluate expression of the p53 gene and induction of apoptosis in tumor and normal tissues exposed to the virus in these patients.
* Evaluate whether transbronchial administration of adenovirus p53 results in improved local tumor control in these patients.

OUTLINE: This is a dose escalation study.

Patients undergo biopsy and receive adenovirus p53 by bronchoalveolar lavage on days 1 and 15. Patients repeat biopsy on days 3 and 28. If there is evidence of clinical benefit or response without significant toxicity, patients may receive a maximum of 3 courses. Treatment beyond 3 courses must be approved by protocol investigator.

Cohorts of 3 patients are treated at escalating dose levels of adenovirus p53. Patients in each cohort are followed for dose limiting toxicity (DLT) for 2 weeks after completion of one course before dose escalation proceeds in subsequent cohorts. If 1 of 3 patients at a dose level experiences dose limiting toxicity (DLT), then 2 additional patients are entered at the same dose level. If more than 1 of 5 patients experience DLT, the previous dose is the maximum tolerated dose (MTD). An additional 10 patients are treated at the MTD.

Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, and annually thereafter.

PROJECTED ACCRUAL: There will be 15 patients accrued into this study over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable non-small cell lung cancer with a growth pattern allowing access to the majority of tumor cells via the airway (e.g., bronchioloalveolar or papillary adenocarcinoma)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Prothrombin time and partial thromboplastin time normal

Hepatic:

* Bilirubin less than 1.5 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* Room air oxygen saturation greater than 90%
* FEV1 greater than 1.0 L pCO2 less than 50

Other:

* HIV negative
* No active systemic viral, bacterial, or fungal infections requiring treatment
* No concurrent illness requiring hospitalization or intravenous medication
* Not pregnant or nursing
* Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior adenovirus gene therapy
* At least 2 weeks since any systemic biologic therapy including prior biologic response modifiers and recovered

Chemotherapy:

* At least 2 weeks since any prior systemic chemotherapy and recovered

Endocrine therapy:

* Recovered from any prior endocrine therapy

Radiotherapy:

* Recovered from any prior radiotherapy

Surgery:

* At least 2 weeks since any surgical procedure requiring anesthesia
* At least 4 weeks since prior surgical resection of lung tissues

Other:

* No other concurrent therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11-17 (Actual); Study Completion 2007-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Carbone, MD, PhD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Result] Keedy V, Wang W, Schiller J, Chada S, Slovis B, Coffee K, Worrell J, Thet LA, Johnson DH, Carbone DP. Phase I study of adenovirus p53 administered by bronchoalveolar lavage in patients with bronchioloalveolar cell lung carcinoma: ECOG 6597. J Clin Oncol. 2008 Sep 1;26(25):4166-71. doi: 10.1200/JCO.2007.15.6927. PMID 18757331
- [Result] Kubba SV, Adak S, Schiller J, et al.: Phase I trial of adenovirus p53 in bronchioalveolar cell lung carcinoma (BAC) administered by bronchioalveolar lavage. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1904, 2000.